CLINICAL TRIAL: NCT00092898
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of Adding Ezetimibe 30 mg to An Ongoing Regimen of Ezetimibe 10 mg in Patients Homozygous Sitosterolemia
Brief Title: An Investigational Drug Study to Lower Non-Cholesterol Sterol Levels Associated With Sitosterolemia (0653-062)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-062; MK0653-062; 2004_038
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Lipid Metabolism, Inborn Errors; Heart Disease
Keywords: Sitosterolemia
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Heart Diseases; Sitosterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: placebo

SUMMARY:
This is a 6-month study with patients who have the rare disease, sitosterolemia which may result in heart-related diseases. These patients have unusually high absorption of non-cholesterol sterols, resulting in heart-related diseases. This study investigates whether absorption of these non-cholesterols can be reduced in these patients.

DETAILED DESCRIPTION:
The duration of treatment is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, with a history of elevated sitosterol levels and have received treatment for at least 6 months prior to study entry.

Exclusion Criteria:

* Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient or interfere with participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2005-09 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Sitosterol concentrations after 26 weeks. | After 26 weeks

SECONDARY OUTCOMES:
Campesterol concentrations; Achilles tendon thickness; safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Musliner T, Cselovszky D, Sirah W, McCrary Sisk C, Sapre A, Salen G, Lutjohann D, von Bergmann K. Efficacy and safety of ezetimibe 40 mg vs. ezetimibe 10 mg in the treatment of patients with homozygous sitosterolaemia. Int J Clin Pract. 2008 Jul;62(7):995-1000. doi: 10.1111/j.1742-1241.2008.01786.x. Epub 2008 May 14. PMID 18484971